CLINICAL TRIAL: NCT02971436
Title: Evaluation of Treatment Efficacy of a Modified Positive Airway Pressure Device to Treat Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: project progression decision was able to be made with the data already gathered
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIA196
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- FPH Device with SensAwake On + Pressure Support A (Active Comparator): FPH Device with SensAwake On + Pressure Support A
  Interventions: Device: FPH Device with SensAwake On + Pressure Support A
- FPH Device with SensAwake Off + Pressure Support A (Active Comparator): FPH Device with SensAwake Off + Pressure Support A
  Interventions: Device: FPH Device with SensAwake Off + Pressure Support A
- FPH Device with SensAwake On + Pressure Support B (Active Comparator): FPH Device with SensAwake On + Pressure Support B
  Interventions: Device: FPH Device with SensAwake On + Pressure Support B
- FPH Device with SensAwake Off + Pressure Support B (Active Comparator): FPH Device with SensAwake Off + Pressure Support B
  Interventions: Device: FPH Device with SensAwake Off + Pressure Support B
- Competitor's PAP Released Device + Pressure Support A (Active Comparator): Competitor's PAP Released Device + Pressure Support A
  Interventions: Device: Competitor's PAP Released Device + Pressure Support A
- Competitor's PAP Released Device + Pressure Support B (Active Comparator): Competitor's PAP Released Device + Pressure Support B
  Interventions: Device: Competitor's PAP Released Device + Pressure Support B

INTERVENTIONS:
Device: FPH Device with SensAwake On + Pressure Support A — FPH Device with SensAwake On + Pressure Support A
  Arms: FPH Device with SensAwake On + Pressure Support A
Device: FPH Device with SensAwake Off + Pressure Support A — FPH Device with SensAwake Off + Pressure Support A
  Arms: FPH Device with SensAwake Off + Pressure Support A
Device: FPH Device with SensAwake On + Pressure Support B — FPH Device with SensAwake On + Pressure Support B
  Arms: FPH Device with SensAwake On + Pressure Support B
Device: FPH Device with SensAwake Off + Pressure Support B — FPH Device with SensAwake Off + Pressure Support B
  Arms: FPH Device with SensAwake Off + Pressure Support B
Device: Competitor's PAP Released Device + Pressure Support A — Competitor's PAP Released Device + Pressure Support A
  Arms: Competitor's PAP Released Device + Pressure Support A
Device: Competitor's PAP Released Device + Pressure Support B — Competitor's PAP Released Device + Pressure Support B
  Arms: Competitor's PAP Released Device + Pressure Support B

SUMMARY:
This study will investigate the efficacy of the FPH modified positive airway pressure (PAP) device with or without SensAwake; and with different pressure support in OSA participants; in both an in-home and in-lab environment. Comfort, compliance and the accuracy of the pressure delivery will also be evaluated. The FPH device will be compared to a market released product.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Diagnosed with OSA by a practicing physician and prescribed Positive Airway Pressure (PAP) - (Continuous Positive Airway Pressure (CPAP) or AutoCPAP). Participants can be naïve to CPAP or experienced users of CPAP.
* For experienced users of PAP (CPAP or AutoCPAP): Using the PAP of more than 4 hours/night for 70% during the last 30 days (justification allowed by the investigator)

Exclusion Criteria:

* Contraindicated for PAP (CPAP or AutoCPAP) therapy
* Persons with other significant sleep disorder(s) (e.g periodic leg movements, insomnia, central sleep apnea)
* Persons with obesity hypoventilation syndrome or congestive heart failure.
* Persons that require supplemental oxygen with their PAP (CPAP or AutoCPAP) device
* Persons with implanted electronic medical device (e.g cardiac pacemakers)
* Persons who are pregnant or think they might be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 3 nights
  Through the device and independent flow logger
Apnea Hypopnea Index (AHI) | 1 night
  Through the polysomnography

SECONDARY OUTCOMES:
Therapy Comfort | 3 nights
  Through a subjective questionnaire
Compliance | 3 nights
  Through the device and independent flow logger
Device Triggering | 3 nights
  Through the device
Device Triggering | 1 night
  Through the polysomnography

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - Fisher & Paykel Healthcare, Auckland
  - WellSleep Centre, Wellington